CLINICAL TRIAL: NCT06745609
Title: Prehabilitation Prior to Surgery for Kidney Tumors: A Randomized Controlled Research Study (Pre-KiT)
Brief Title: Prehabilitation Prior to Surgery for Kidney Tumors
Acronym: Pre-KiT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Herlev and Gentofte Hospital (Other)
Responsible Party: Principal Investigator, Marie Mykløy Haslund, M.D., PhD-student, Herlev and Gentofte Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: H-24066449
Record Dates: First submitted 2024-12-12; First posted 2024-12-20 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Renal Cancer; Renal Cell Cancer; Kidney Cancers; Stage I Renal Cell Cancer; Prehabilitation; Elderly (People Aged 65 or More)
Keywords: Prehabilitation; Quality of life; Kidney tumor; Renal cell tumor; Renal cell cancer; Kidney cancer; Quality of recovery; Elderly
MeSH Terms: conditions — Kidney Neoplasms; Carcinoma, Renal Cell | interventions — Preoperative Exercise; Geriatric Assessment; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (No Intervention): Participants in the control group are scheduled for surgery in compliance with the Danish cancer patient pathway guarantees (within 14 days).
- Intervention with Pre-KiT prehabilitation (Experimental): Participants in the intervention group are scheduled for surgery after four weeks of Pre-KiT prehabilitation. The prehabilitation consists of a geriatric guided assessment with relevant targeted interventions, a home exercise program and assisted smoking cessation.
  Interventions: Other: Prehabilitation

INTERVENTIONS:
Other: Prehabilitation — Pre-KiT prehabilitation consists of
  1. A geriatric guided assessment with relevant interventions. The assessment will include cognitive evaluation, screening for depression, functional assessment, as well as evaluation of nutritional risk, assessment of past and current diseases, and a thorough review of the patient's medication list focusing on drug interactions. It will also include social history and standard laboratory results,
  2. Physical activity. A four week home exercise program, adjusted to the participants physical abilities.
  3. Assisted smoking cessation
  Other Names: Geriatric assessment; Physical activity; Smoking cessation
  Arms: Intervention with Pre-KiT prehabilitation

SUMMARY:
The goal of this clinical trial is to examine if one month of general health optimization before surgery for kidney tumors can help participants recover more quickly from surgery.

The optimization process is called prehabiliation, and will last one month. It consists of

1. A comprehensive health assessment
2. Assisted smoking cessation
3. A home exercise program.

The investigators will compare an intervention group receiving one month of prehabilitation with a control group receiving the standard of care.

Some of the main questions the investigators want to answer are

* Are participants in the intervention group more satisfied with their quality of recovery after surgery?
* Do participants in the intervention group maintain more of their physical abilites compared to the control group?

ELIGIBILITY:
Inclusion Criteria:

* 65 years or older
* cT1 kidney tumor, scheduled for either partial or radical nephrectomy.
* Clinical Frailty Scale 3-6

Exclusion Criteria:

* It is determined by an attending physician, or at a multi-disciplinary team-conference, that a 2-4 week postponement of surgery will not be beneficial for the participant.
* Participant does not understand Danish og English

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-01-21 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2032-03 (Estimated)

PRIMARY OUTCOMES:
Change in quality of recovery from screening to outpatient follow-up 21 days after surgery | From enrollment to outpatient follow-up at 21 days after surgery.
  Quality of recovery is evaluated with the danish translation of the verified questionnaire Quality of Recovery-15. It is a 15-item patient questionnaire, where the score ranges from 0-150. A higher score indicates better patient-reported quality of recovery. QoR-15 will be assessed at enrollment, preoperatively, and 1, 21 and 90 days after surgery. Change in QoR-15 from enrollment to 21 days after surgery is the primary outcome measure. Change in QoR-15 at other assessment times will be assessed as secondary outcome measures.

SECONDARY OUTCOMES:
Change in Quality of Recovery at other times | Multiple times from enrollment to outpatient follow-up at 90 days after surgery.
  Quality of recovery is measured by the danish translation of the verified questionnaire Quality of Recovery-15. It is a 15-item patient questionnaire, where the score ranges from 0-150. A higher score indicates better patient-reported quality of recovery. QoR-15 will be assessed at enrollment, preoperatively, and 1, 21 and 90 days after surgery.
Change in the 30 second chair stand test | Multiple times from enrollment to outpatient follow-up at 90 days after surgery.
  Physical ability is measured by the 30 second chair stand test. The test is performed at enrollment, preoperatively, 21 and 90 days after surgery.
Change in hand grip strength | Multiple times from enrollment to outpatient follow-up at 90 days after surgery.
  Physical ability is measured by hand grip strength. The test is performed with a hand-dynamometer at enrollment, preoperatively, 21 and 90 days after surgery.
Compliance to the prehabilitation program | From enrollment to the preoperative assessment
  Compliance to the prehabilitation program is measured by brief phone interviews with the study participants in the intervention group two times a week during the intervention.
Days alive and out of hospital 90 days | From hospital discharge to follow-up 90 days after surgery.
  Days alive and out of hospital (DAOH) is the number of days not in hospital after surgery. DAOH will be calculated at 90 days after surgery.
Change in Quality of Life | Multiple times from enrollment to outpatient follow-up at 90 days after surgery.
  Quality of life is evaluated with the danish translation of the validated questionnaire EQ-5D-5L. The questionnaire evalutes five health dimensions (mobility, self-care, usual acitivites, pain/discomfort, anxiety/depression) ranging from "no problems" to "unable/ extreme problems". Additionally, it includes a visual analog scale scoring from 0-100, reflecting the participants overall self-reported health state. A higher score indicates a better patient-reported quality of life. Quality of life will be assessed at enrollment, preoperatively, 21 and 90 days after surgery.
Medical and surgical complications defined according to Clavien-Dindo at 30 and 90 days after surgery | At 30 and 90 days after surgery.
  Clavien-Dindo is a system to summarize and classify postoperative complications. Complications will be identified in participants records, and scored according to the Clavien-Dindo grades I-V, where V is the most severe. Registration of complications will be conducted at 30 and 90 days after surgery.
Health economic analysis | From enrollment to 1 year follow-up
  Health-related expenses associated with standard treatment and PreKiT-based treatment will be analyzed and compared across the two study arms.
Survival | From surgery to 5 year follow-up.
  Recurrence-free survival, Cause-specific survival and overall survival measured at 1 and 5 years after surgery.
Change in muscle mass | From enrollment to 1 year follow-up
  Change in muscle mass, comparing measures on preoperative-CT and one year follow-up CT, including assessment of sarcopenia according to current European guidelines.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Urology, Herlev and Gentofte Hospital, Herlev, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Juul-Haslund M, Lund CM, Dolin TG, Schou-Jensen K, Ostergren PB, Vinther A, Thomsen FF, Fode M. Geriatric prehabilitation prior to surgery for kidney tumors: Study protocol for Pre-KiT - A randomized controlled trial. J Geriatr Oncol. 2026 Jan 26;17(2):102893. doi: 10.1016/j.jgo.2026.102893. Online ahead of print. PMID 41592385